CLINICAL TRIAL: NCT06515002
Title: A Seamless Phase I/II Trial With an Initial Open-label Dose Escalation Part and a Subsequent Randomised, Double-blind, Placebo-controlled Expansion Part to Evaluate the Safety, Tolerability, and Efficacy of a Single Dose of BI 3720931, an Inhaled Lentiviral Vector Gene Therapy, in Adult People With Cystic Fibrosis Who Are Ineligible for CFTR Modulators (Lenticlair 1)
Brief Title: A Study to Test How Well BI 3720931 is Tolerated and Whether it Improves Lung Function in People With Cystic Fibrosis (Lenticlair™ 1)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1504-0001; 2023-503281-23-00 (Registry Identifier: CTIS); U1111-1291-0800 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP)); 1504.1 (Other: Sponsor ID)
Record Dates: First submitted 2024-07-18; First posted 2024-07-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Intervention Model Description: The open-label dose escalation part, Phase I, will study the safety and efficacy of single doses of three different dose levels of BI 3720931 in trial participants with cystic fibrosis (CF).
  Phase II will be a double-blind, placebo-controlled, dose expansion part with 3 arms: first arm investigating Phase II dose 1, second arm investigating Phase II dose 2, and third arm for placebo.
  An interim analysis of the safety and efficacy data from Phase I will be used for the decision making to move to Phase II and the selection of doses in Phase II.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phase I: open-label Phase II: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Phase I: Dose group 1 (low dose) (Experimental)
  Interventions: Genetic: BI 3720931; Device: Inhaler
- Phase I: Dose group 2 (medium dose) (Experimental)
  Interventions: Genetic: BI 3720931; Device: Inhaler
- Phase I: Dose group 3 (high dose) (Experimental)
  Interventions: Genetic: BI 3720931; Device: Inhaler
- Phase II: Dose group 1 (Experimental)
  Interventions: Genetic: BI 3720931; Device: Inhaler
- Phase II: Dose group 2 (Experimental)
  Interventions: Genetic: BI 3720931; Device: Inhaler
- Phase II: Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo; Device: Inhaler

INTERVENTIONS:
Genetic: BI 3720931 — BI 3720931
  Arms: Phase I: Dose group 1 (low dose); Phase I: Dose group 2 (medium dose); Phase I: Dose group 3 (high dose); Phase II: Dose group 1; Phase II: Dose group 2
Drug: Placebo — Placebo
  Arms: Phase II: Placebo group
Device: Inhaler — Inhaler for application of BI 3720931 and placebo

SUMMARY:
This study is open to adult men with cystic fibrosis and adult women with cystic fibrosis who cannot have children. People with cystic fibrosis can join if they are not eligible to receive cystic fibrosis transmembrane conductance regulator modulator therapy (CFTR-MT). The purpose of this study is to find out how well a medicine called BI 3720931 is tolerated and whether it improves lung function in people with cystic fibrosis. In this study, BI 3720931 is given to humans for the first time.

This study has two phases. In Phase 1, participants are put in one of 3 groups, one group after the other. Each group gets a different dose of BI 3720931. Group 1 starts with the lowest dose, followed by group 2 with the middle and group 3 with the high dose. In Phase 2, participants are put into 3 groups by chance, but at the same time. 2 groups get different doses of BI 3720931 selected based on results of Phase 1, and 1 group gets placebo. All study participants get only 1 dose of BI 3720931 or placebo and they use a special inhaler to take the study medicine. The placebo inhaler looks like the BI 3720931 inhaler but does not contain any medicine. During the study, participants continue taking their usual medicines.

Doctors closely monitor participants' health at the study site for the first 3 days after receiving BI 3720931. Participants visit their doctors regularly thereafter. The doctors check the health of the participants and note any health problems that could have been caused by BI 3720931. Study participants regularly do a standard lung function test to measure how well their lungs are working. Participants, in either Phase 1 or Phase 2, are in the study for 7 months. After completion of this study, participants will take part in a long-term follow-up study (1504-0003).

ELIGIBILITY:
Key inclusion criteria:

* Cystic fibrosis (CF)-pulmonary phenotype and a confirmed diagnosis of CF:

  * Positive sweat chloride ≥60 mmol/L by pilocarpine iontophoresis OR
  * Genotype with 2 identifiable CF-causing mutations accompanied by one or more clinical features if sweat chloride testing is between 30 and 59 mmol/L
* Trial participants who are not eligible for treatment with cystic fibrosis transmembrane conductance regulator modulator therapy (CFTRmt) due to their genotype with 2 identified CFTR-mutations (including Class I CFTR gene mutations) and are also not expected to become eligible during the trial according to investigator´s opinion
* Trial participants able to perform acceptable spirometric maneuvers according to American Thoracic Society/European Respiratory Society 2019 standards
* Forced expiratory volume in 1 second, percent of predicted value (FEV1pp) ≥50% and ≤100% of predicted normal at Visit 1. Predicted value based on Global Lung Initiative lung function reference equations
* Stable CF disease with no pulmonary exacerbation 4 weeks prior to the screening visit and during the screening period and stable drug- and non-drug therapy for CF in the 4 weeks prior to dosing Further inclusion criteria apply.

Key exclusion criteria:

* Trial participants not eligible for CFTRmt based on contraindications (e.g. liver failure) or who needed to withdraw CFTRmt due to intolerability are not appropriate candidates for this Phase I/II trial
* Trial participants requiring chronic use of systemic corticosteroids or immunosuppressants to treat another condition Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2028-03-14 (Estimated); Study Completion 2028-07-04 (Estimated)

PRIMARY OUTCOMES:
Phase I: Occurrence of any drug-related, treatment-emergent adverse events (AE) up to Week 24 after drug administration | up to 24 weeks
Phase II: Absolute change from baseline in forced expiratory volume in 1 second, percent of predicted value (FEV1pp) at Week 8 after drug administration | at baseline, at week 8

SECONDARY OUTCOMES:
Phase I: Occurrence of treatment response defined as change from baseline ≥5% in FEV1pp, comparing the mean of 3 pre-treatment FEV1pp measured in the screening period with the mean of 3 post-treatment FEV1pp-values at Weeks 4, 6, and 8 | up to 12 weeks
Phase I: Absolute change from baseline in FEV1pp at Week 24 after drug administration | at baseline, at week 24
Phase I: Occurrence of any dose limiting toxicities (DLTs) up to Week 24 after drug administration | up to 24 weeks
Phase II: Absolute change from baseline in FEV1pp at Week 24 after drug administration | at baseline, at week 24
Phase II: Occurrence of any serious adverse events (SAEs) up to Week 24 after drug administration | up to 24 weeks
Phase II: Occurrence of any drug-related, treatment-emergent AEs up to Week 24 after drug administration | up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- France (2):
  - HOP Gui de Chauliac, Montpellier
  - HOP Necker, Paris
- Italy (2):
  - Istituto G. Gaslini, Genova
  - Osp. Pediatrico Bambin Gesù, Roma
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Hospital Universitari Vall D Hebron, Barcelona, Spain
- United Kingdom (4):
  - University Hospital Llandough, Cardiff
  - Queen Elizabeth University Hospital, Glasgow
  - Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com